CLINICAL TRIAL: NCT03549520
Title: Improved Diagnosis and Prognostication of Hypoxic Ischemic Injury in Neonates and Infants Using Contrast-Enhanced Ultrasound
Brief Title: CEUS Evaluation of Hypoxic Ischemic Injury
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Bracco Diagnostics, Inc (Industry)
Responsible Party: Principal Investigator, Misun Hwang, MD, Sponsor Investigator, Children's Hospital of Philadelphia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-014912
Record Dates: First submitted 2018-05-25; First posted 2018-06-08 (Actual); Results first posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Hypoxic-Ischemic Encephalopathy; Brain Ischemia Hypoxia
Keywords: Ultrasound; Contrast-enhanced ultrasound
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Contrast-enhanced Ultrasonography (Experimental): Intravenous administration of contrast agent Sulfur hexafluoride lipid-type A microspheres before performing contrast-enhanced ultrasound (CEUS). In pediatric patients, after reconstitution 0.03 mL per kg is administered intravenously. The weight-based dose of 0.03 mL per kg will be repeated one time during a single examination. Following each injection, an intravenous flush of 0.9% Sodium Chloride is injected. The study duration per subject will be approximately 15 minutes including the time to prepare the contrast agent and perform the CEUS, as well as the 60 minute monitoring period after the first and second injection of the contrast agent.
  Interventions: Drug: Sulfur hexafluoride lipid-type A microspheres

INTERVENTIONS:
Drug: Sulfur hexafluoride lipid-type A microspheres — Injection of Sulfur hexafluoride lipid-type A microspheres (Lumason) contrast agent will be performed via the existing peripheral intravenous line using the FDA-recommended dose of 0.03 mg/kg.

SUMMARY:
Neonates presenting with neurologic symptoms require rapid, non-invasive imaging with high spatial resolution and tissue contrast. The purpose of this study is to evaluate brain perfusion using contrast-enhanced ultrasound CEUS in bedside monitoring of neonates and infants with hypoxic ischemic injury (HII). Investigational CEUS scan will be performed separately from clinically indicated conventional US, in the ICU. Subjects will be scanned with CEUS at two different time-points (at the time HII is first suspected or diagnosed and at time of MRI scan), separately from clinically indicated ultrasound. The CEUS scan will be interpreted by the sponsor-investigator.

The study will be conducted at one site, The Children's Hospital of Philadelphia. It is expected that up to 100 subjects will be enrolled per year, for up to two years, for a total enrollment of up to 200 subjects.

DETAILED DESCRIPTION:
Contrast-enhanced ultrasonography (CEUS) is a novel imaging technique in which gas-filled microbubbles, smaller than red blood cells, generate increased signal due to the acoustic impedance mismatch. Injection of ultrasound contrast agents into blood increase the echogenicity, allowing enhanced visualization of a blood vessel. Ultrasound contrast agents have been approved for use in Europe for almost two decades. In the case of SonoVue (now called LumasonTM), a second-generation lipid/sulfur hexafluoride US contrast agent (Bracco, Milan, Italy), European Union approved its intravenous use in adults in 2001. The FDA in the United States just recently approved the use of LumasonTM for evaluation of focal hepatic lesions in pediatric population in 2016, and very recently (Jan 2017) approved its use in children for the evaluation of the urinary tract in pediatric patients with known or suspected vesicoureteral reflux. For the remainder of clinical applications, the ultrasound contrast agents are being used off-label in both Europe and the United States.

There is already good evidence in the literature that CEUS may be very valuable in children, and that is why it is routinely performed off-label for this purpose in the USA. However, there are ways in which it could be improved, and more studies are needed to definitively establish its diagnostic performance.

Sulfur hexafluoride lipid-type A microspheres (LumasonTM, Bracco Inc) is an FDA-approved ultrasound contrast agent. The study duration per subject will be approximately 15 minutes including the time to prepare LumasonTM contrast agent and perform the CEUS, as well as the 60 minute monitoring period after the first and second injection of LumasonTM. CEUS will be performed at the time HII is first suspected or diagnosed and within 24 hours of clinically indicated MRI (which occurs approximately on day 5 of life) for a total of two CEUS exams of 1 hour and 15-minute duration each. Study participation will be complete when the 60 minute monitoring period after the second CEUS is complete.

Injection of LumasonTM contrast agent will be performed via the existing peripheral intravenous line or central line using the FDA-recommended dose of up to 0.03 mg/kg. Contrast-agent injection will be performed twice per CEUS scan to ensure image quality and test reproducibility. In the case of more stable patients without an IV line, a peripheral IV line will be started to conduct the investigational CEUS. Two bolus injections will performed to evaluate for dynamic brain perfusion and several 2-minute cine clips as well as static images will be acquired during the exam.

Qualitative analysis with visual assessment and quantitative analysis of the acquired CEUS scans will be performed and interpreted by the PI. The scans will be assessed for diagnostic quality of images, artifacts encountered, and the presence of additional contributory diagnostic information.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 1.5 years or younger with open fontanelles and known or suspected hypoxic ischemic injury.
2. Post menstrual age of 34 weeks or older
3. Patient in the Children's Hospital of Philadelphia (CHOP) Neonatal Intensive Care Unit (NICU) or Pediatric Intensive Care Unit (PICU)
4. Parental permission

Exclusion Criteria:

1. Medical history of Lumason hypersensitivity
2. Hemodynamic instability as defined by rapid escalation of cardiopulmonary support in the past 12-24 hours, as defined by the clinical care team including ≥ 1 intensive care physician not part of the study team
3. Pulmonary insufficiency as defined by fraction of inspired oxygen (FiO2) requirements of > 40% and/or subjects with pulmonary hypertension requiring nitric oxide

Ages: 1 Minute to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hwang M, Piskunowicz M, Darge K. Advanced Ultrasound Techniques for Pediatric Imaging. Pediatrics. 2019 Mar;143(3):e20182609. doi: 10.1542/peds.2018-2609. PMID 30808770

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Main reasons for lack of enrollment were the presence of clinical instability and/or pulmonary insufficiency/hypertension.
Groups:
- Brain Contrast-enhanced Ultrasonography: Intravenous administration of contrast agent Sulfur hexafluoride lipid-type A microspheres before performing contrast-enhanced ultrasound (CEUS). In pediatric patients, after reconstitution 0.03 mL per kg is administered intravenously. The weight-based dose of 0.03 mL per kg will be repeated one time during a single examination. Following each injection, an intravenous flush of 0.9% Sodium Chloride is injected. The study duration per subject will be approximately 15 minutes including the time to prepare the contrast agent and perform the CEUS, as well as the 60 minute monitoring period after the first and second injection of the contrast agent.
Period: Overall Study
Arm/Group | Brain Contrast-enhanced Ultrasonography
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Low enrollment. Main reason was not fulfillment of inclusion/exclusion criteria, either for clinical instability and/or pulmonary insufficiency/hypertension.
Groups:
- Brain Contrast-enhanced Ultrasonography: Intravenous administration of contrast agent Sulfur hexafluoride lipid-type A microspheres before performing contrast-enhanced ultrasound (CEUS). In pediatric patients, after reconstitution 0.03 mL per kg is administered intravenously. The weight-based dose of 0.03 mL per kg will be repeated one time during a single examination. Following each injection, an intravenous flush of 0.9% Sodium Chloride is injected. The study duration per subject will be approximately 15 minutes including the time to prepare the contrast agent and perform the CEUS, as well as the 60 minute monitoring period after the first and second injection of the contrast agent.
  Sulfur hexafluoride lipid-type A microspheres: Injection of Sulfur hexafluoride lipid-type A microspheres (Lumason) contrast agent will be performed via the existing peripheral intravenous line using the FDA-recommended dose of 0.03 mg/kg.
Arm/Group | Brain Contrast-enhanced Ultrasonography
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Days] | 14 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Detection of Brain Perfusion Abnormalities Using Contrast-enhanced Ultrasound
Description: Comparison of brain perfusion between normal subjects (those with suspected or at risk of HII but turn out to be normal on imaging and clinical evaluation) versus HII patients
Time Frame: During contrast-enhanced ultrasound examination, up to 15 minutes.
Population: One subject was enrolled, therefore, no comparison was possible. The patient presented with HII confirmed by MRI.
Measure: Number; unit: Participants
Groups:
- Brain Contrast-enhanced Ultrasonography: Intravenous administration of contrast agent Sulfur hexafluoride lipid-type A microspheres before performing CEUS through an existing peripheral intravenous line using the FDA-recommended dose of 0.03 mg/kg. Two bolus injections will be performed and several 2-minute cine clips as well as static images will be acquired during the exam.
Arm/Group | Brain Contrast-enhanced Ultrasonography
Number analyzed (Participants) | 1
Participants
  Patients with HII who underwent CEUS examination | 1
  Patients without HII who underwent CEUS examination | 0

2. Secondary Outcome: Number of Participants With Completed Brain CEUS Exams, Categorized by Diagnostic-Quality Scoring System
Description: Scoring system of non-diagnostic (1), moderate artifacts degrading diagnostic quality (2), mild artifacts without degradation of diagnostic quality (3), and diagnostic (4).
Time Frame: During contrast-enhanced ultrasound examination, up to 15 minutes.
Population: Evaluation of brain CEUS diagnostic quality
Measure: Number; unit: Participants
Arm/Group | Brain Contrast-enhanced Ultrasonography
Number analyzed (Participants) | 1
Participants
  Non-diagnostic | 0
  Mild artifacts without degradation of diagnostic quality | 0
  Moderate artifacts degrading diagnostic quality | 0
  Diagnostic | 1

ADVERSE EVENTS:
Time Frame: 15 Minutes.
Arm/Group | Brain Contrast-enhanced Ultrasonography
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/20/NCT03549520/Prot_SAP_000.pdf